CLINICAL TRIAL: NCT05891860
Title: Virtual Family Participation in ICU Rounds (The VR-Family Study)
Brief Title: Virtual Family Participation in ICU Rounds: a Pilot Study
Acronym: VR-Family
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Davis Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Fonds de la Recherche en Santé du Québec (Other Government); McGill Faculty of Medicine (Unknown)
Responsible Party: Principal Investigator, Michael Goldfarb, Attending Staff, Division of Cardiology, Lady Davis Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023-3581
Record Dates: First submitted 2023-03-20; First posted 2023-06-07 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Family Engagement; Virtual; Critical Care
Keywords: family engagement; virtual; critical care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Study participants will be present during daily ICU team rounds by secure video conference.
  Interventions: Other: Participation in virtual rounds

INTERVENTIONS:
Other: Participation in virtual rounds — Virtual participation in daily ICU team rounds

SUMMARY:
Barriers to family participation in ICU rounds exist at the health care system level (e.g., restriction on visitation, infection control) and the individual level (e.g., caretaker role, illness, disability, inability to miss work). While virtual family participation in ICU rounds may contribute to addressing these barriers, its feasibility, impact, and effectiveness are yet unknown. The primary objective of this study is to assess the feasibility of virtual family participation in adult ICU rounds. The secondary objectives are: to assess the effect size of virtual family participation in ICU rounds on family engagement, satisfaction, and anxiety and depression; and to explore family and physician experiences of family participation in ICU rounds.

This will be a pilot prospective trial of 72 family members at 4 Canadian adult ICUs, with an embedded qualitative study that will sample family members and critical care physicians. The primary outcome will reflect feasibility metrics (i.e., recruitment, uptake, technical, and follow-up). Secondary outcomes include data regarding family engagement, satisfaction, mental health, and perceived experiences of participation in ICU rounds. This study will assess the feasibility of conducting a larger, hypothesis-testing randomized controlled trial to assess virtual family participation in adult ICU rounds.

ELIGIBILITY:
Inclusion Criteria:

* Family member of ICU patient with expected ICU stay > 48 hours (as per treating team)
* Age ≥ 18 years old
* Willing and able to participate in virtual ICU rounds
* Ability to communicate in English or French
* Able: technological capability and understanding to participate virtually in ICU rounds (must have a phone or computer with internet and audio/video capabilities).
* "Family member" is anyone with a biological, legal, or emotional relationship with the patient.

Exclusion criteria

* Intends to participate in in-person rounds (if available and offered at participating site)
* Another family member already participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Recruitment rate of 3 participants per month per site completing initial FAME questionnaire | 6 months
  Recruitment rate
% of participants completing at least one virtual rounding session | Within 1-week of ICU discharge
  Uptake
% of virtual rounds without technical issues | Within 1-week of ICU discharge
  Technical issues
% of participants completing follow-up | Within 1-week of ICU discharge
  Follow-up of participants

SECONDARY OUTCOMES:
Family satisfaction as measured by FS-ICU 24R | Within 1-week of ICU discharge
  Family satisfaction
Anxiety and depression as measured by HADS | Within 1-week of ICU discharge
  Anxiety and depression
Family care engagement as measured by FAME | Within 1-week of ICU discharge
  Family care engagement

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calderone A, Debay V, Goldfarb MJ. Family Presence on Rounds in Adult Critical Care: A Scoping Review. Crit Care Explor. 2022 Nov 7;4(11):e0787. doi: 10.1097/CCE.0000000000000787. eCollection 2022 Nov. PMID 36382337
- [Background] Au SS, Roze des Ordons AL, Blades KG, Stelfox HT. Best practices toolkit for family participation in ICU rounds. J Eval Clin Pract. 2021 Oct;27(5):1066-1075. doi: 10.1111/jep.13517. Epub 2020 Nov 23. PMID 33230927
- [Background] Davidson JE, Aslakson RA, Long AC, Puntillo KA, Kross EK, Hart J, Cox CE, Wunsch H, Wickline MA, Nunnally ME, Netzer G, Kentish-Barnes N, Sprung CL, Hartog CS, Coombs M, Gerritsen RT, Hopkins RO, Franck LS, Skrobik Y, Kon AA, Scruth EA, Harvey MA, Lewis-Newby M, White DB, Swoboda SM, Cooke CR, Levy MM, Azoulay E, Curtis JR. Guidelines for Family-Centered Care in the Neonatal, Pediatric, and Adult ICU. Crit Care Med. 2017 Jan;45(1):103-128. doi: 10.1097/CCM.0000000000002169. PMID 27984278